CLINICAL TRIAL: NCT05034107
Title: Effects of Diffused Ylang-Ylang (Cananga Odorata) Essential Oil Amongst Older Persons With Dementia: A Pre-Post Quasi-Experimental Study Protocol
Brief Title: Effects of Diffused Ylang-Ylang Essential Oil Amongst Older Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Collaborators: Universiti Sains Malaysia (Other); University of Malaya (Other)
Responsible Party: Principal Investigator, Shubashini Gnanasan, Principal Investigator, Universiti Teknologi Mara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FRGS/1/2017/SKK02/UITM/02/1
Record Dates: First submitted 2021-08-22; First posted 2021-09-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Dementia; Behavioral and Psychiatric Symptoms of Dementia
Keywords: Aromatherapy; Ylang-Ylang; Behavioral and Psychological Symptoms of Dementia; Dementia
MeSH Terms: conditions — Dementia; Behavior | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: A pre-post quasi-experimental study will be conducted over a two-month period in nursing homes with persons with dementia. During the pre-intervention phase, essential oil diffusers containing water will be diffused in the common area of the nursing homes. During the intervention phase, Ylang-Ylang essential oil will be diffused using an identical diffuser. Behavioural parameters and blood samples will be taken after pre and post intervention phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persons with dementia (Experimental): Persons who have been diagnosed with dementia by their physicians and in nursing homes. Persons with dementia who have at least one symptom of BPSD and willing to participate in this study. These participants will be exposed to diffused Ylang-Ylang aromatherapy.
  Interventions: Other: Aromatherapy

INTERVENTIONS:
Other: Aromatherapy — Approximately 6-7 drops of Ylang-ylang essential oil will be diffused in a common area estimated to be about 300 square feet with temperature of around 25 - 26 degree Celsius and humidity of 50% - 60%. Water and essential oil will be diffused twice a day, each for a duration of 20 min during the respective phases.
  Other Names: Ylang-Ylang; Young Living® Essential Oils (Ylang-Ylang)

SUMMARY:
Ylang-Ylang (Cananga Odorata) essential oil has been postulated to have calming effect, which may improve BPSD in persons with dementia. This study aims to examine dementia-related behavioural changes using established assessment tools and brain derived neurotropic factor (BDNF) in persons with BPSD.

DETAILED DESCRIPTION:
Behavioural and Psychological Symptoms of Dementia (BPSD) refers to the spectrum of non-cognitive and non-neurological symptoms of dementia, such as agitation, psychosis, depression and apathy. Ylang-Ylang (Cananga Odorata) essential oil is postulated to have calming effect, which may improve BPSD in persons with dementia. Thus, this study aims to examine dementia-related behavioural changes using established assessment tools and brain derived neurotropic factor (BDNF) in persons with BPSD. A pre-post quasi-experimental pilot study will be conducted over a two-month period in nursing homes with persons with dementia. Approximately 30 persons with dementia are expected to participate in this study. During the pre-intervention phase, water will be diffused using a diffuser in a common area of the nursing homes. During the intervention phase, Ylang-Ylang essential oil will be diffused using the identical diffuser over the same common area. Both water and essential oil will be diffused twice a day, each for a duration of 20 min during the respective phases. Observation and documentation of behavioural symptoms will be taken using validated instruments during the pre- and post-intervention phases. In addition, 10 mL of blood will also be collected at pre and post intervention for biochemical analyses.If Ylang-ylang essential oil were found to be beneficial based on the laboratory and observational findings, it can be possibly used as an alternative approach in managing BPSD.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have been diagnosed with dementia by their physicians and in nursing homes in Selangor, Malaysia.
* Persons with dementia who have at least one symptom of BPSD

Exclusion Criteria:

* Persons with dementia with a comorbid respiratory problem like asthma or chronic obstructive pulmonary disease
* Persons with dementia who are allergic to fragrance/perfumes
* Persons with dementia who had a change in their psychotropic or dementia medications in the 30 days before commencement of the study, namely: acetylcholinesterase inhibitors N-methyl-D-aspartate (NMDA)-receptor antagonist (memantine), antipsychotics, antidepressants, sedatives, or medications with anticholinergic properties
* Persons who have been diagnosed with schizophrenia or mental retardation
* Persons who have no documented behavioral history in the previous three month
* Persons who are currently hospitalized
* Persons with dementia who are unwilling to participate or disallowed by caregivers/family members

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Cornell Scale for Depression in Dementia | 2 months
  The mean counts of this parameter before and after intervention phase will be analysed using Cornell Scale for Depression in Dementia. The score more than 18 means the persons is having definite major depressive episode.
Cohen-Mansfield Agitation Inventory | 2 months
  The mean counts of this parameter before and after the intervention phase will be analysed using Cohen-Mansfield Agitation Inventory. A rating of five indicates that the person is having frequent agitation within an hour.
Neuropsychiatric Inventory- Brief Questionnaire Form | 2 months
  The mean counts of this parameter before and after the intervention phase will be analysed using the Neuropsychiatric Inventory- Brief Questionnaire Form. A person is undergoing severe symptoms of BPSD if the score is 3, while caregivers are undergoing more distress when the score is 5.

SECONDARY OUTCOMES:
Serum BDNF (100μL) | 2 months
  Enzyme linked immunosorbent assay (ELISA) will be used.
Amyloid Beta (Aβ1-40) (100μL) | 2 months
  Enzyme linked immunosorbent assay (ELISA) will be used.
Amyloid Beta (Aβ1-42) (100μL) | 2 months
  Enzyme linked immunosorbent assay (ELISA) will be used.
cytokines (150μL ) | 2 months
  IL-2, IL-6, IL-8, and TNF-α levels will be tested using Plex Proteomic Assay kit.
Cortisol( 50μL) | 2 months
  Enzyme linked immunosorbent assay (ELISA) will be used.
adrenocorticotropic hormone (50μL) | 2 months
  Enzyme linked immunosorbent assay (ELISA) will be used.
MDA(Malondialdehyde) (50μL) | 2 months
  Enzyme linked immunosorbent assay (ELISA) will be used.
Reduced Glutathione (GSH) (0.7 mL) | 2 months
  Colorimetric Assay Kit will be used.
Thiobarbituric Acid Reactants (TBARS) (0.1mL) | 2 months
  Colorimetric Assay Kit will be used.
Total Antioxidant Capacity (T-AOC) (10 μL) | 2 months
  Colorimetric Assay Kit will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Shubashini Gnanasan, PhD, Principal Investigator — Universiti Teknologi Mara
Locations (1):
- Universiti Teknologi MARA, Kuala Selangor, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No